CLINICAL TRIAL: NCT02153281
Title: Neuroimaging MAO-B in Medication Free and Treatment Resistant Major Depressive Disorder Using Novel MAO-B Tracer
Brief Title: Neuroimaging MAO-B in Medication Free TR-MDD Using Novel Tracer
Acronym: DETB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Jeff Meyer, Head Neurochemical Imaging in Mood Disorders, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DETB-071-13
Record Dates: First submitted 2014-03-28; First posted 2014-06-03 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Positron Emission Tomography (PET); MAO-B
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phenelzine treatment (Experimental): Subjects will undergo a PET and MRI scan before and after the treatment.
  Interventions: Other: phenelzine treatment

INTERVENTIONS:
Other: phenelzine treatment — Subjects will have a PET and MRI scan before and after treatment with phenelzine.

SUMMARY:
The purpose of this study is to determine if monoamine oxidase B (MAO-B) total distribution volume (VT), after phenelzine treatment and if so to what extent.

DETAILED DESCRIPTION:
Subjects will receive a PET and MRI scan before and after treatment with phenelzine.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* good physical health
* Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) diagnosis of current major depressive episode (MDE)
* DSM-IV diagnosis of major depressive disorder (MDD) verified by SCID for DSM-IV and a psychiatric consultation
* greater than 17 on the 17 item HDRS (Hamilton Depression Rating Scale).
* history of non-response to several different antidepressant classes

Exclusion Criteria:

* herbal, drug or medication use (that affect CNS function)
* suicide attempts
* drug or medication use within eight weeks (+5 half lives of medication)
* history of substance abuse or any neurotoxin use
* history of psychotic symptoms
* history of central nervous system (CNS) medical illness
* current substance abuse
* test positive on pregnancy test (for women)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-06; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
MAO-B VT levels measured with PET in MDE secondary to MDD | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H. Meyer, MD, PhD, Principal Investigator — Research Imaging Centre, Centre for Addiction and Mental Health
Locations (1):
- Center for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/research